CLINICAL TRIAL: NCT04412603
Title: Conventional Mirror Therapy and Mirror Therapy Virtual Reality in Obstetric Brachial Palsy: Pilot Study
Brief Title: Emergent Therapies in OBP. Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Obstetric Brachial Palsy
Record Dates: First submitted 2020-02-19; First posted 2020-06-02 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Neonatal Brachial Plexus Palsy
Keywords: Virtual Reality.; family; Mirror Therapy; Obstetrical Brachial Palsy; Upper extremity
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy

STUDY DESIGN:
Intervention Model Description: A pilot randomized clinical trial was performed with simple blind and randomization of block assignmen.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Mirror Therapy group (Experimental): Therapy:
  -With the affected upper limb into the mirror box, perform the exercise with the non-affected extremity which is reflected in the mirror box. -The affected side must perform the corresponding movement within its possibilities, according to the exercise that is being performed with the healthy arm. - It is very important to look at the mirror at all times, which reflects the non-affected side while doing the exercises.
  Interventions: Other: Conventional Mirror Therapy
- Mirror Therapy Virtual Reality group (Experimental): Therapy:
  -Perform the exercises with the non-affected limb, which must be watched constantly with virtual reality glasses, to interpret that this limb corresponds to the affected side. - The affected side accompanies the movement within its possibilities (out of sight of the patient, it can be covered with a handkerchief). - It is very important to look at the non-affected side. The affected side should be out of the visual field to avoid confusion.
  Interventions: Other: Conventional Mirror Therapy

INTERVENTIONS:
Other: Conventional Mirror Therapy — The Conventional Mirror Therapy was carried out with a mirror box and the Mirror Therapy Virtual Reality was carried out with virtual reality glasses and mobile application: Mirror Therapy VR.
  Other Names: Mirror Therapy Virtual Reality

SUMMARY:
Obstetric Brachial Palsy (OBP) produces functional limitations in the involvement of the affected upper limb within the child's natural environment. The therapeutic interventions of Conventional Mirror Therapy (MT) and Mirror Therapy Virtual Reality (VR) are aimed at the rehabilitation of the affected upper limb and the quality life improvement.

To quantify the increase in the affected upper limb spontaneous use and the quality of life of children with upper OBP from 6-12 years, when They are treated with Conventional MT or Mirror Therapy VR applying specific protocol: 20 min/day in 4 weeks.

DETAILED DESCRIPTION:
The intervention protocol was permorfed for four weeks, three days per week applying Conventional Mirror Therapy or Mirror Therapy Virtual Reality, with 20-minute sessions in 4 weeks. Designed to be done at home.

Two measurements of the affected upper limb spontaneous use and quality of life were performed, a pre-treatment assessment corresponding to the baseline situation, and another post-treatment Assessment to observe the results after the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 6 and 12 years old, upper Obstetric Brachial Palsy type Erb-Duchenne (C5-C6) and extended Erb-Duchenne (C5-C7), preserved functionality to do the activities, adequate cognitive level to follow the proposed activities.

Exclusion Criteria:

* associated pathologies, medical complications or cognitive and / or visual impairment that prevent the activities performance, affected upper limb surgeries in the last year, treatment with botulinum toxin in the last three months, no possession of a device with Android operating system for the application of Virtual Reality therapy, families and children no partners.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Children's Hand-use Experience Questionnaire | Four weeks
  To measure the affected upper limb spontaneous use, validated for children with unilateral involvement or disuse of one of their upper limbs from 6 to 18 years in which the experience of children using the affectected upper limb.
Pediatric Quality of Life Inventory Generic Core Scales PedsQLTM 4.0 | Four weeks
  Modular instrument for measuring health-related quality of life in children and adolescents ages 2 to 18.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Palomo, Physiotherapist, Study Director — San Pablo-CEU Univerity
Locations (1):
- San Pablo-CEU Univerity, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No